CLINICAL TRIAL: NCT05425407
Title: A Randomized Double-blinded Placebo-controlled Study to Evaluate the Effect of Collagen Peptide (Collagen Peptan) Supplementation on Muscle and Tendon Damage, Repair, and Functional Capacity During Exercise Training Overload
Brief Title: Effects of Collagen Peptide Supplementation on Muscle and Tendon Damage and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Rousselot BVBA (Industry)
Responsible Party: Principal Investigator, Peter Hespel, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S64402
Record Dates: First submitted 2021-08-03; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Exercise; Healthy Male Subjects
Keywords: Whey protein; Collagen peptide; Muscle and tendon overload training
MeSH Terms: conditions — Motor Activity | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Only whey protein will be provided
  Interventions: Dietary Supplement: whey protein
- Collagen (Experimental): A mix of whey protein and collagen peptides will be provided
  Interventions: Dietary Supplement: whey protein + collagen peptide

INTERVENTIONS:
Dietary Supplement: whey protein — Daily 45g of whey protein supplementation during a three week eccentric training period
  Arms: Placebo
Dietary Supplement: whey protein + collagen peptide — Daily 15g of whey protein and 20g collagen peptide supplementation during a three week eccentric training period
  Arms: Collagen

SUMMARY:
The aim of the study is to investigate the acute and short-term effects of collagen peptides (Collagen Peptan) on muscle and connective tissue during an eccentric overload training period. Currently, all studies investigating the effects of post-exercise collagen supplementation did this in the absence of whey proteins, which are part of the standard recommendations for post-exercise recovery. The investigators will therefore investigate whether the combined intake of whey proteins and collagen peptides ensures a better recovery of exercise performance and whether it can prevent or reduce symptoms of muscle and tendon overload during a three-week eccentric overload training period (n = 22).

ELIGIBILITY:
Inclusion Criteria:

* Sports participation, including general fitness training, between 2 and 5 hours max per week
* Body mass index between 18.5 and 25

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform high-intensity exercise - Intake of any medication or nutritional supplement that could impact muscle protein synthesis and/or exercise performance during the period of the study
* Intake of any whey protein, casein of branched-chain amino acid (BCAA) supplements from 1 month prior to the start of the study
* Blood donation within 3 months prior to the start of the study
* Smoking
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in countermovement jump performance | Pretest - 48 hours after the first training session (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Change in jump height when performing a countermovement jump, measured via a force platform
Change in maximal isometric knee-extension force of the right leg | Pretest - 48 hours after the first training session (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Change in maximal isometric knee-extension force (angle = 45°) of the right leg
Change in anteroposterior thickness of the right patellar tendon | Pretest - 48 hours after the first training session (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Change in anteroposterior thickness of the right patellar tendon
Change in neovascularization of the right patellar tendon | Pretest - 48 hours after the first training session (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Neovascularization of the right patellar tendon scored with the Modified Ohberg Score (range 0 - 4; the higher the score, the higher the degree of neovascularization).

SECONDARY OUTCOMES:
Change in pain perception at the muscular level (VAS scale) | Training 1 (day 1 of training intervention) - Training 2 (day 3 of training intervention) - Training 8 (day 9 of training intervention) - Training 17 (day 19 of training intervention) - Posttest (day 22 of training intervention)
  Change in pain perception at the muscular level of the right leg, measured via the Visual Analogue Scale (range 0 - 10; the higher the score, the higher the pain level)
Change in pain perception of the patellar tendon of the right leg (VISA-P) | Pretest - Training 1 (day 1 of training intervention) - Training 17 (day 21 of training intervention) - Posttest (day 22 of training intervention)
  Change in pain perception of the patellar tendon of the right leg, measured via the VISA-P questionnaire (range: 0 - 100; the lower the score, the higher the symptoms of patellar tendon overload)
Change in the blood concentration of creatine kinase | Pretest - Training 2 (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Change in blood concentration of creatine kinase (marker of muscle damage)
Change in the blood concentration of Interleukin 6 (IL-6) | Pretest - Training 2 (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Change in blood concentration of Interleukin 6 (IL-6; marker of inflammation)
Change in the blood concentration of N-terminal propeptide of type I procollagen (P1NP) | Pretest - Training 2 (day 3 of training intervention) - Posttest (day 22 of training intervention)
  Change in blood concentration of N-terminal propeptide of type I procollagen (P1NP; marker of collagen synthesis)

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Research Group, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided